CLINICAL TRIAL: NCT06216444
Title: A Multi-center, Randomized, Double-blind Clinical Study to Evaluate the Efficacy and Safety of Remimazolam Tosilate (Ruibeining®) for Injection for Sedation in Non-intubated Diagnostic and Therapeutic Procedures
Brief Title: A Study of Remimazolam Tosilate for Sedation in Non-intubated Diagnostic and Therapeutic Procedures
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HR7056-401
Record Dates: First submitted 2023-12-27; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Sedation in Non-intubated Diagnostic and Therapeutic Procedures
MeSH Terms: interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam Tosilate for Injection（5mg） (Experimental)
  Interventions: Drug: Remimazolam Tosilate for Injection
- Remimazolam Tosilate for Injection（10mg） (Experimental)
  Interventions: Drug: Remimazolam Tosilate for Injection

INTERVENTIONS:
Drug: Remimazolam Tosilate for Injection — Initial loading dose of 5mg, with additional doses of 2.5mg as necessary
  Arms: Remimazolam Tosilate for Injection（5mg）
Drug: Remimazolam Tosilate for Injection — Initial loading dose of 10mg, with additional doses of 2.5mg as necessary
  Arms: Remimazolam Tosilate for Injection（10mg）

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Remimazolam Tosilate for Injection for sedation in non-intubated diagnostic and therapeutic procedures

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, male or female
2. Intending to undergo routine gastroscopy or colonoscopy
3. ASA (American Society of Anesthesiologists) I to III
4. 18 kg/m2≤BMI (Body Mass Index)≤30kg/m2
5. Signed informed consent

Exclusion Criteria:

1. Subjects need to be tracheal intubation
2. Subjects need to be complicated endoscopic diagnostic and therapeutic procedures
3. Subjects who have had severe cardiovascular diseases or severe arrhythmias within 6 months prior to signing the ICF
4. Heart rate <50 beats/min during the screening period
5. Poor blood pressure control during the screening period
6. Subjects with severe respiratory diseases
7. Subjects with respiratory management difficulties (Modified Mallampati grade IV)
8. Subjects with a history of mental illness (schizophrenia, mania, bipolar disorder, psychosis, etc.), long-term use of psychotropic drugs, and cognitive impairment
9. A history of drug abuse or addiction within 2 years prior to signing the ICF
10. Pregnant women or those in lactation period
11. Allergic to relevant drugs ingredient or component in the study
12. Currently participating in or planning to participate in other drug or device clinical trials during this study
13. Other conditions deemed unsuitable to be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Rate of sedation success, Sedation success | day 1
  Rate of sedation success, Sedation success is defined as: 1) Completion of the entire non-intubated diagnostic and therapeutic procedure; 2) No need for additional rescue sedation; 3) During the sedation induction phase, the MOAA/S score should be ≤3 within 2 minutes after the end of the initial dose administration or after ≤2 additional administrations; 4) No more than 2 additional administrations in every 5-minute.

SECONDARY OUTCOMES:
Number of additional administrations. | day 1
Percentage of subjects needing additional administration. | day 1
One-time success rate of endoscope insertion during the diagnostic and therapeutic procedure. | day 1
Rate of over-sedation. | day 1
Sedation induction time | day 1
Wake-up time. | day 1
Time to discharge. | day 1
Rate of sedation-related hypotension and rate of sedation-related hypotension needing treatment. | day 1
Rate of respiratory depression during sedation. | day 1
Investigator's Satisfaction with Sedation Assessment: The scoring range is from 0 to 10, where 0 represents dissatisfaction and 10 represents complete satisfaction. | day 1
Participant's satisfaction with Sedation Assessment: The scoring range is from 0 to 10, where 0 represents dissatisfaction and 10 represents complete satisfaction. | day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided